CLINICAL TRIAL: NCT06551181
Title: A Phase 3, Randomized, Controlled, Partially Blind, Immuno-bridging Study to Evaluate Immunogenicity, Reactogenicity, Safety and the Occurrence of RSV Associated Respiratory Tract Illness After Administration of a Single Dose of GSK's RSVPreF3 OA Investigational Vaccine in Adults Aged 60 Years and Older
Brief Title: A Study on the Immune Response, Safety and the Occurrence of Respiratory Syncytial Virus (RSV)-Associated Respiratory Tract Illness After Administration of RSV OA Vaccine in Adults 60 Years and Older
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 219815; 2023-509455-13-00 (Other: EU CTR Number)
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Respiratory syncytial virus (RSV); Older adults; Acute respiratory illness (ARI); Lower respiratory tract disease (LRTD); Immune response; Efficacy study; Safety study
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Data from study participants in China is collected in an observer-blind manner. The study is open labelled for overseas participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RSV OA vaccine Group (China) (Experimental): Chinese participants receive a single dose of RSVPreF3 OA investigational vaccine at Day 1 and are followed up until end of study (Month 6 or last ARI visit/contact, whichever is later).
  Interventions: Biological: RSVPreF3 OA investigational vaccine
- Placebo Group (China) (Placebo Comparator): Chinese participants receive a single dose of placebo at Day 1 and are followed up until end of study (Month 6 or last ARI visit/contact, whichever is later).
  Interventions: Drug: Placebo
- RSV OA vaccine Group (Overseas) (Experimental): Overseas participants receive a single dose of RSVPreF3 OA investigational vaccine at Day 1 and are followed up until end of study (Month 6).
  Interventions: Biological: RSVPreF3 OA investigational vaccine

INTERVENTIONS:
Biological: RSVPreF3 OA investigational vaccine — One dose of the RSVPreF3 OA investigational vaccine is administered intramuscularly at Day 1.
  Arms: RSV OA vaccine Group (China); RSV OA vaccine Group (Overseas)
Drug: Placebo — One dose of placebo is administered intramuscularly at Day 1.
  Arms: Placebo Group (China)

SUMMARY:
The purpose of the current study is to evaluate the immune response of the RSVPreF3 OA investigational vaccine in older adults (OA) at least (>=) 60 years of age (YOA) in China compared to OA in the same age range to be enrolled from overseas countries that participated in the RSV OA=ADJ-006 (NCT04886596) study, since the vaccine efficacy against lower respiratory tract disease (LRTD) has been demonstrated following a single dose of the RSVPreF3 OA investigational vaccine in the global efficacy study RSV OA=ADJ-006. In addition, the safety (in all participants) , reactogenicity and occurrence of RSV-associated acute respiratory illness (ARI) (in study participants in China only) after administration of the vaccine are also assessed in the current study. No ARI surveillance will be conducted for the overseas participants.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female of ≥60 YOA at the time of study intervention administration, who live in the community dwelling (CD participants).
* Participants who, in the opinion of the investigator, can and will comply with the requirements of the protocol (e.g., completion of the diary cards, attend regular phone calls/study site visits, perform self-swabbing (study participants in China only), ability to access and utilize a phone or other electronic communications).
* Participants who are medically stable in the opinion of the investigator at the time of vaccination. Participants with chronic stable medical conditions with or without specific treatment, such as diabetes, hypertension or cardiac disease, are allowed to participate in this study if considered by the investigator as medically stable.
* Written or witnessed informed consent obtained from the participant (participant must be able to understand the informed consent) prior to performance of any study specific procedure.

Exclusion Criteria:

Medical Conditions:

* History of any reaction or hypersensitivity likely to be exacerbated by any component of the study intervention(s).
* Any clinical conditions for which serum samples would be prohibited for transfer to local central lab for testing. These clinical conditions include hepatitis B, hepatitis C, HIV and Syphilis based on medical history and physical examination (all participants) and laboratory screening tests (overseas participants).
* Any confirmed or suspected immunosuppressive or immunodeficient condition resulting from disease (e.g., current malignancy, human immunodeficiency virus) or immunosuppressive/cytotoxic therapy (e.g., medication used during cancer chemotherapy, organ transplantation, or to treat autoimmune disorders), based on medical history and physical examination (no laboratory testing required).
* Any history of dementia or any medical condition that moderately or severely impairs cognition.
* Recurrent history or uncontrolled neurological disorders or seizures. Participants with medically controlled active or chronic neurological diseases can be enrolled in the study as per investigator assessment, provided that their condition will allow them to comply with the requirements of the protocol (e.g. completion of the diary cards, attend regular phone calls/study site visits, perform self-swabbing (study participants in China only).
* Significant underlying illness that in the opinion of the investigator would be expected to prevent completion of the study (e.g., life-threatening disease likely to limit survival to less than 1 year).
* Serious or unstable chronic illness.
* Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the participant due to participation in the study.

Prior/Concomitant Therapy:

* Previous vaccination with RSV vaccine.
* Use of any investigational or non-registered product (drug, vaccine or invasive medical device) other than the study intervention(s) during the period beginning 30 days before the dose of study intervention(s), or their planned use during the study period.
* Planned or actual administration of a vaccine not foreseen by the study protocol in the period starting 30 days before and ending 30 days after study intervention administration, with the exception of COVID-19 and inactivated/subunit influenza vaccines which can be administered up to 14 days before or from 14 days after each study intervention.
* Administration of long-acting immune-modifying drugs or planned administration at any time during the study period (e.g., infliximab).
* Administration of immunoglobulins and/or any blood products or plasma derivatives during the period starting 90 days before the study intervention administration or planned administration during the study period.
* Chronic administration (defined as more than 14 consecutive days in total) of immunosuppressants or other immune-modifying drugs during the period starting 90 days prior to the study intervention administration or planned administration during the study period. For corticosteroids, this will mean prednisone >=20 mg/day, or equivalent. Inhaled and topical steroids are allowed.

Prior/Concurrent Clinical Study Experience:

• Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational intervention (drug/invasive medical device).

Other Exclusion Criteria:

* History of chronic alcohol consumption and/or drug abuse as deemed by the investigator to render the potential participant unable/unlikely to provide accurate safety reports or comply with study procedures.
* Bedridden participants.
* Planned move during the study conduct that prohibits participation until study end.
* Participation of any study personnel or their immediate dependents, family, or household members.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2621 (Actual)
Dates: Start 2024-08-05 (Actual); Primary Completion 2025-04-24 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
RSV-A neutralization titers expressed as geometric mean titers (GMTs) in RSV OA vaccine Group (Overseas) and RSV OA vaccine Group (China), and between-group GMT ratios | At 1 month after the RSVPreF3 OA investigational vaccine administration (Day 31)
  RSV-A neutralization titers are determined by neutralization assay and expressed as GMTs.
Percentage of participants showing group seroresponse for RSV-A in RSV OA vaccine Group (Overseas) and RSV OA vaccine Group (China), and between-group differences | At 1 month after the RSVPreF3 OA investigational vaccine administration (Day 31)
  A participant with seroresponse for RSV-A is defined as a participant having at least a 4-fold increase in RSV-A neutralizing titers (1 month post-study intervention administration over pre-study intervention administration >=4).
RSV-B neutralization titers expressed as geometric mean titers (GMTs) in RSV OA vaccine Group (Overseas) and RSV OA vaccine Group (China), and between-group GMT ratios) | At 1 month after the RSVPreF3 OA investigational vaccine administration (Day 31)
  RSV-B neutralization titers are determined by neutralization assay and expressed as GMTs.
Percentage of participants showing group seroresponse for RSV-B in RSV OA vaccine Group (Overseas) and RSV OA vaccine Group (China), and between-group differences | At 1 month after the RSVPreF3 OA investigational vaccine administration (Day 31)
  A participant with seroresponse for RSV-B is defined as a participant having at least a 4-fold increase in RSV-B neutralizing titers (1 month post-study intervention administration over pre-study intervention administration >=4).

SECONDARY OUTCOMES:
RSV-A neutralization titers expressed as GMTs in RSV OA vaccine Group (Overseas) and RSV OA vaccine Group (China) | At Baseline (Day 1), at 1 month (Day 31) and at 6 months (Day 181) after the RSVPreF3 OA investigational vaccine administration
RSV-B neutralization titres expressed as GMTs in RSV OA vaccine Group (Overseas) and RSV OA vaccine Group (China) | At Baseline (Day 1), at 1 month (Day 31) and at 6 months (Day 181) after the RSVPreF3 OA investigational vaccine administration
Percentage of participants showing seroresponse for RSV-A in RSV OA vaccine Group (Overseas) and RSV OA vaccine Group (China) | At 1 month (Day 31) and at 6 months (Day 181) after the RSVPreF3 OA investigational vaccine administration
  A participant with seroresponse for RSV-A is defined as a participant having at least a 4-fold increase in RSV-A neutralizing titers (1 month post-study intervention administration over pre-study intervention administration >=4).
Percentage of participants showing seroresponse for RSV-B in RSV OA vaccine Group (Overseas) and RSV OA vaccine Group (China) | At 1 month (Day 31) and at 6 months (Day 181) after the RSVPreF3 OA investigational vaccine administration
  A participant with seroresponse for RSV-B is defined as a participant having at least a 4-fold increase in RSV-B neutralizing titers (1 month post-study intervention administration over pre-study intervention administration >=4).
RSV-A neutralization titers expressed as group GMTs in the immunogenicity subset of RSV OA=ADJ-006 study and in RSV OA vaccine Group (China) | At 1 month after the RSVPreF3 OA investigational vaccine administration (Day 31)
RSV-B neutralization titers expressed as group GMTs in the immunogenicity subset of RSV OA=ADJ-006 study and in RSV OA vaccine Group (China) | At 1 month after the RSVPreF3 OA investigational vaccine administration (Day 31)
Percentage of participants showing seroresponse for RSV-A in the immunogenicity subset of RSV OA=ADJ-006 study and in RSV OA vaccine Group (China) | At 1 month after the RSVPreF3 OA investigational vaccine administration (Day 31)
  A participant with seroresponse for RSV-A is defined as a participant having at least a 4-fold increase in RSV-A neutralizing titers (1 month post-study intervention administration over pre-study intervention administration >=4).
Percentage of participants showing seroresponse for RSV-B in the immunogenicity subset of RSV OA=ADJ-006 study and in RSV OA vaccine Group (China) | At 1 month after the RSVPreF3 OA investigational vaccine administration (Day 31)
  A participant with seroresponse for RSV-B is defined as a participant having at least a 4-fold increase in RSV-B neutralizing titers (1 month post-study intervention administration over pre-study intervention administration >=4)
Number of participants with real time polymerase chain reaction (RT-PCR) confirmed RSV-A associated ARI and LRTD in RSV OA vaccine Group (China) and Placebo Group (China) | From the RSVPreF3 OA investigational vaccine administration (Day 1) to Month 6
  ARI is characterized by the presence of at least 2 respiratory symptoms/signs for at least 24 hours OR at least 1 respiratory symptom/sign + 1 systemic symptom/sign for at least 24 hours. An RT-PCR-confirmed RSV-ARI is defined as an event meeting the case definition of ARI with at least one RSV-positive swab detected by RT-PCR. LRTD is characterized by the presence of at least 2 lower respiratory symptoms/signs for at least 24 hours including at least 1 lower respiratory sign OR at least 3 lower respiratory symptoms for at least 24 hours. An RT-PCR-confirmed RSV-LRTD is defined as an event meeting the case definition of LRTD with at least one RSV-positive swab . detected by RT-PCR.
Number of participants with RT-PCR confirmed RSV-B associated ARI and LRTD RSV OA vaccine Group (China) and Placebo Group (China) | From the RSVPreF3 OA investigational vaccine administration (Day 1) to Month 6
  ARI is characterized by the presence of at least 2 respiratory symptoms/signs for at least 24 hours OR at least 1 respiratory symptom/sign + 1 systemic symptom/sign for at least 24 hours. An RT-PCR-confirmed RSV-ARI is defined as an event meeting the case definition of ARI with at least one RSV-positive swab detected by RT-PCR. LRTD is characterized by the presence of at least 2 lower respiratory symptoms/signs for at least 24 hours including at least 1 lower respiratory sign OR at least 3 lower respiratory symptoms for at least 24 hours. An RT-PCR-confirmed RSV-LRTD is defined as an event meeting the case definition of LRTD with at least one RSV-positive swab . detected by RT-PCR.
Number of participants with solicited administration site events in RSV OA Group (China) and Placebo Group (China) | Within 7 days after study intervention administration (the day of study intervention administration and the subsequent 6 days)
  The assessed solicited administration site events are pain, erythema and swelling.
Number of participants with solicited systemic events in RSV OA Group (China) and Placebo Group (China) | Within 7 days after study interventions (the day of study intervention administration and the subsequent 6 days)
  The assessed solicited systemic events are fever, headache, myalgia, arthralgia and fatigue.
Number of participants with unsolicited adverse events (AEs) in RSV OA Group (China) and Placebo Group (China) | Within 30 days after study interventions (the day of study intervention administration and the subsequent 29 days)
  An unsolicited AE is an AE that was either not included in the list of solicited events or could be included in the list of solicited events but with an onset outside the specified period of follow-up for solicited events. Unsolicited AEs must have been communicated by participants who has signed the informed consent.
Number of participants with serious adverse events (SAEs) in all study groups | From the study intervention administration (Day 1) to Month 6
  An SAE is defined as any untoward medical occurrence that results in death, are life threatening, require hospitalization or prolongation of hospitalization or results in disability/incapacity.
Number of participants with potential immune-mediated disease (pIMDs) in all study groups | From the study intervention administration (Day 1) to Month 6
  pIMDs are a subset of Adverse Events of Specific Interest (AESIs) that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology.
Number of participants with SAEs related to study intervention in all study groups | From the study intervention administration (Day 1) to study end (approximately 6 months post dose administration)
  An SAE is defined as any untoward medical occurrence that results in death, are life threatening, require hospitalization or prolongation of hospitalization or results in disability/incapacity.
Number of participants with pIMDs related to study interventions in all study groups | From the RSVPreF3 OA investigational vaccine administration (Day 1) to study end (approximately 6 months post dose administration)
  pIMDs are a subset of Adverse Events of Specific Interest (AESIs) that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology.
Number of participants with any fatal SAEs in all study groups | From the RSVPreF3 OA investigational vaccine administration (Day 1) to study end (approximately 6 months post dose administration)
  An SAE is defined as any untoward medical occurrence that results in death, are life threatening, require hospitalization or prolongation of hospitalization or results in disability/incapacity.

CONTACTS AND LOCATIONS:
Locations (35):
- China (3):
  - GSK Investigational Site, Shanghai, Putuo
  - GSK Investigational Site, Shanghai, Shanghai Municipality
  - GSK Investigational Site, Shanghai
- Finland (7):
  - GSK Investigational Site, Espoo
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Kokkola
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Seinäjoki
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
- GSK Investigational Site, Tokyo, Japan
- Poland (8):
  - GSK Investigational Site, Elblag
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Sochaczew
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wroclaw
- South Korea (3):
  - GSK Investigational Site, Guri-si
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Seoul
- Spain (6):
  - GSK Investigational Site, Ávila
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Burgos
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Salamanca
  - GSK Investigational Site, Valladolid
- United Kingdom (7):
  - GSK Investigational Site, Belfast
  - GSK Investigational Site, Blackpool
  - GSK Investigational Site, Bristol
  - GSK Investigational Site, Cambridgeshire
  - GSK Investigational Site, Eynsham
  - GSK Investigational Site, Hounslow
  - GSK Investigational Site, Witney

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/